CLINICAL TRIAL: NCT06243783
Title: Impact of Acute Stress and Its Habituation on Brain Energy Metabolism
Brief Title: Impact of Stress on Brain Energy Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rupert Lanzenberger (Other)
Collaborators: University of Konstanz (Other)
Responsible Party: Sponsor-Investigator, Rupert Lanzenberger, Prof. PD MD, Head Neuroimaging Labs, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSY-NIL-0012
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress (Experimental): Montreal Imaging Stress Test during each PET/MRI measurement and in-between
  Interventions: Behavioral: Montreal Imaging Stress Test

INTERVENTIONS:
Behavioral: Montreal Imaging Stress Test — In the Montreal Imaging Stress Test, participants are required to solve basic mathematical tasks, but the allowed reaction time is set lower than their average.

SUMMARY:
Background: Stress plays an essential role in the pathophysiology of mental disorders. However, individual differences in the vulnerability to acute and repeated stress are not well understood.

Aim: This work aims to investigate individual differences in glucose metabolism and directional connectivity regulating the neuronal stress response.

Design: 68 healthy volunteers will undergo two simultaneous PET/MRI measurements one week apart. Participants will complete the Montreal Imaging Stress Test during each measurement and in-between. Effects of stress on cognitive performance will be assessed using the n-back working memory task. Individual cortisol levels will be acquired to identify stress (non)responders as well as (non)habituators.

Implications: This work will characterize differences between stress responders vs. non-responders and stress habituators vs. non-habituators in terms of energy metabolism and network connectivity. This individual difference in the stress response may represent an important cornerstone for future evaluation of patients with mental disorders.

DETAILED DESCRIPTION:
Methodological details: Each participant will undergo two PET/MRI scans. Imaging will include functional PET and as well as structural and functional MRI. Stress-specific glucose metabolism will be quantified with the radioligand [18F]FDG. Functional connectivity will be combined with glucose metabolism to assess directional connectivity. Based on previous literature, changes are expected to occur in the anterior cingulate cortex.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* right-handedness
* willingness and competence to sign the informed consent form

Exclusion Criteria:

* History of or current physical, neurological or psychiatric disorder
* History of or current substance abuse or medication, including antipsychotic, antidepressant and antianxiety agents
* Pregnancy of current breast-feeding
* Contraindications for MRI-scanning (e.g., metal implants, steel grafts, etc.), including dental implants causing signal artifacts
* For subjects participating in earlier studies using ionizing radiation, the total radiation exposure of 30 mSv over the last 10 years must not be exceeded, as specified in the Austrian legislation on radiation protection Accordingly, body weight > 105 kg is an exclusion criterion.
* Failure to comply with the study protocol or to follow the instructions of the investigating team.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Stress induced changes in glucose metabolism | 1 week
  Glucose metabolism will be quantified from [18F]FDG PET imaging.

SECONDARY OUTCOMES:
Stress induced changes in directional connectivity | 1 week
  Directional connectivity will be computed as combination of MRI-based functional connectivity and glucose metabolism.
Stress induced changes in cognitive performance | 1 week
  Cognitive performance will be obtained by the n-back working memory task.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hahn, Assoc.Prof., Principal Investigator — Department of Psychiatry and Psychtherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be deposited on datadryad.
Time Frame: After study completion.
Access Criteria: Public access.

REFERENCES:
- See also: Neuroimaging Labs, Dept. of Psychiatry and Psychotherapy, Medical University of Vienna — https://www.meduniwien.ac.at/neuroimaging/